CLINICAL TRIAL: NCT04539275
Title: VA CoronavirUs Research and Efficacy Studies-1 (VA CURES-1)
Brief Title: VA CoronavirUs Research and Efficacy Studies-1
Acronym: VACURES-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: DMC recommended early termination of enrollment
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COVID19-8900-22
Record Dates: First submitted 2020-08-27; First posted 2020-09-04 (Actual); Results first posted 2022-09-10 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: COVID-19
Keywords: 2019 novel coronavirus disease; COVID-19 pandemic; COVID-19 virus infection; COVID-19 virus disease; Respiratory failure; Pneumonia, viral / therapy; Blood Component Transfusion; Severity of Illness Index; Survival Analysis; Treatment Outcome; Prospective Study; Humans; Adults; Male; Female; convalescent plasma; SARS CoV-2; COVID-19 convalescent plasma
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency; Pneumonia | interventions — COVID-19 Serotherapy; Saline Solution

STUDY DESIGN:
Intervention Model Description: There are two study treatment arms: convalescent plasma versus saline. Participants will be randomized in 1:1 ratio to these two arms.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The participants, site investigators, clinical prescribers, site coordinators, and most other individuals involved in this study will be blinded to the treatment assignment.
  Furthermore, the blind will not routinely be broken in order to select post-study, pharmacologic treatment for SARS-CoV-2 infection administered by clinical healthcare providers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Convalescent Plasma (Experimental): The study intervention consists of intravenous administration of 200-500 mL of convalescent plasma administered in two equally divided doses, less than 12 hours apart.
  Interventions: Drug: Convalescent Plasma
- Masked Saline Placebo (Placebo Comparator): The study intervention consists of intravenous administration of 200-500 mL of 0.9% saline administered in two equally divided doses, less than 12 hours apart.
  Interventions: Other: Masked Saline Placebo

INTERVENTIONS:
Drug: Convalescent Plasma — Convalescent plasma from persons recovered from SARS-CoV-2 is being used to treat hospitalized individuals with complicated COVID-19 infection.
  Other Names: COVID-19 Convalescent Plasma (CCP)
  Arms: Convalescent Plasma
Other: Masked Saline Placebo — 0.9% saline solution will be used as the Masked Saline Placebo
  Other Names: Normal Saline (NS)
  Arms: Masked Saline Placebo

SUMMARY:
The purpose of this study is to determine if treatment with convalescent plasma improves the clinical outcomes of Veterans who are hospitalized and require supplemental oxygen due to COVID-19.

DETAILED DESCRIPTION:
As of August 25, 2020, SARS-Coronavirus 2 (SARS-CoV-2; COVID-19) infections are approaching 6 million persons and 180,000 deaths in the US. Of the 20% of patients admitted to hospital, up to half progress to ICU admission, respiratory failure or death. Prominent among these progressors are older men, particularly those with underlying comorbidities (e.g., hypertension, diabetes, lung, heart, kidney or liver disease, obesity and immunocompromised), all common among Veterans. There are no drugs or other therapeutics approved by the FDA to prevent or treat COVID-19 infection.

Convalescent plasma therapy is being used empirically, although only five of six small uncontrolled case series (total n=56) in SARS-CoV-23-8 and a recent study with non-randomized controls suggest improved selected clinical, virologic and laboratory outcomes; outcomes in another small randomized trial were equivocal. For other infections, such as influenza and Ebola virus, promising observational studies were not reliably confirmed by controlled trials. In multiple infections, use of convalescent plasma has been distinguished by its safety profile but not by the consistency of its benefit.

The current double-blind, placebo-controlled randomized clinical trial (RCT) is designed to determine definitively whether this intervention is effective in a population at high risk of complications and death from SARS-CoV-2 infection. The investigators compare the effect of convalescent plasma vs. saline placebo with a robust study design, adequate sample size and statistical and logistical rigor to assure that the interventions the investigators make to treat serious disease are well-validated to support its use or to move on to test other potentially safe and effective treatments.

This study is taking place at approximately 25 Veterans Affairs (VA) Medical Centers located across the US. A participant's involvement will last up to 33 days. The entire study, from the date the first person enters until the last participant is seen, is expected to last about 20 months.

Data collected for this study will be analyzed and stored at the Palo Alto Cooperative Studies Program Coordinating Center (CSPCC). After the study is completed, the de-identified, archived data will continue to be stored at the Palo Alto CSPCC, accessible for use by researchers including those outside of the study with an approved Data Use Agreement. The biospecimens collected in the study for current and future research will be kept at the VA Biorepository in Palo Alto, California unless otherwise specified. The biospecimens will be accessible for future research with an approved Sample Use Agreement. The VA Central Institutional Review Board (CIRB) will oversee the biorepository for this study. All samples will be destroyed by standard practice within 20 years of study completion. Sample destruction will be validated according to the Standard Operating Procedures of the VA Biorepository.

ELIGIBILITY:
Inclusion Criteria:

Veterans must meet all of the following criteria to be eligible to participate:

1. Admitted to a participating VA clinical site with symptoms suggestive of SARS-CoV-2 infection.
2. Participant (or legally authorized representative) provides informed consent prior to initiation of any study procedures.
3. Participant (or legally authorized representative) understands and agrees to comply with planned study procedures.
4. Veteran 18 years of age at time of screening.
5. Has laboratory-confirmed SARS-CoV-2 infection as determined by polymerase chain reaction (PCR) or antigen test, as documented by either of the following:

(1)Reverse Transcription polymerase chain reaction (RT-PCR) or antigen positive (nasopharyngeal, oropharyngeal, saliva, lower respiratory) in sample collected 72 hours prior to screening; (2)RT-PCR or antigen positive in sample collected > 72 hours but 168 hours (i.e. 7 days) prior to screening, documented inability to obtain a repeat sample (e.g. due to lack of testing supplies, limited testing capacity, results taking > 24 hours, etc.), AND progressive disease suggestive of ongoing SARS-CoV-2 infection.

6.Requiring oxygen by nasal cannula or by face-mask as a new treatment (or if previously on home oxygen, at a liter flow at least 2 Lpm greater than home prescription), but not on humidified heated high-flow nasal cannula (HHHFNC) at 15 Lpm.

7.Can be randomized within 72 hours of hospital admission. 8.Agrees not to participate in another therapeutic clinical trial for the treatment of COVID-19 or SARS-CoV-2 through Day 29 without approval from the investigator(s). Taking part in other research studies, including those unrelated to SARS-CoV-2, without first discussing it with the investigators of this study may invalidate the results of this study, as well as that of the other study.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Respiratory failure requiring mechanical ventilation, non-invasive ventilation including continuous positive airway pressure (CPAP) (for an indication other than previously diagnosed sleep apnea and maintained on outpatient settings), or extra-corporeal membrane oxygenation or anticipated to require any of those treatments or to die within 24 hours.
2. Anticipated discharge from the hospital or transfer to another hospital that is not a study site within 72 hours.
3. History of previous transfusion reaction.
4. Previously documented serum immunoglobulin A (IgA) deficiency (<7 mg/dL)
5. Documented to have received convalescent plasma in the last 60 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward N. Janoff, MD, Study Chair — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (24):
- United States (23):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Orlando VA Medical Center, Orlando, FL, Orlando, Florida
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan
  - VA Southern Nevada Healthcare System, North Las Vegas, NV, North Las Vegas, Nevada
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Oklahoma City VA Medical Center, Oklahoma City, OK, Oklahoma City, Oklahoma
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin
- VA Caribbean Healthcare System, San Juan, PR, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Janoff EN, Shih MC, Donskey C, Belitskaya-Levy I, Brau N, Rodriguez-Barradas MC, Chan E, Zimmerman P, Miller EK, Vaughan LB, Daniel Markley J, Goldberg AM, Sriram P, Anzueto A, Uyeda L, Zehm L, Wills A, Hutchinson C, Jones L, Peterson D, Ringer RJ, Dumont L, Gleason T, Bonomo RA, Curtis JL, Brown ST; CURES-1 Trials Consortium. Impact of High-Titer Convalescent Plasma on Clinical and Virologic Outcomes Among Veterans Hospitalized With SARS-CoV-2 Infection: VA CoronavirUs Research and Efficacy Studies-1 (VA CURES-1). J Med Virol. 2025 May;97(5):e70349. doi: 10.1002/jmv.70349. PMID 40400480
- [Derived] Janoff EN, Brown ST, Belitskaya-Levy I, Curtis JL, Bonomo RA, Miller EK, Goldberg AM, Zehm L, Wills A, Hutchinson C, Dumont LJ, Gleason T, Shih MC; ADD Caitlin MS in CCTC website. Design of VA CoronavirUs Research and Efficacy Studies-1 (VA CURES-1): A double-blind, randomized placebo-controlled trial of COVID-19 convalescent plasma in hospitalized patients with early respiratory compromise. Contemp Clin Trials Commun. 2023 Jul 17;35:101190. doi: 10.1016/j.conctc.2023.101190. eCollection 2023 Oct. PMID 37560085
- [Derived] Miller EK, Goldberg AM, Janoff EN, Brown ST, Curtis JL, Bonomo RA, Shih MC, Gleason TC. Designing and implementing methodology for double-blind, placebo-controlled clinical trials using blood products within the Department of Veterans Affairs. Clin Trials. 2022 Apr;19(2):137-145. doi: 10.1177/17407745211069703. Epub 2022 Mar 1. PMID 35229691

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Convalescent Plasma | Masked Saline Placebo
Started | 35 | 40
Received Study Product | 32 | 40
Completed | 29 | 35
Not Completed | 6 | 5
Not completed — Death | 2 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Convalescent Plasma | Masked Saline Placebo | Total
Number analyzed (Participants) | 35 | 40 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 18 | 34
  >=65 years | 19 | 22 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (14.5) | 67 (11.5) | 66.4 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 34 | 38 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 17
  Not Hispanic or Latino | 26 | 31 | 57
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 15 | 26
  White | 21 | 22 | 43
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 40 | 75
Clinical Status [Count of Participants; unit: Participants]
  Ambulatory, no limitation of activity | 0 | 0 | 0
  Ambulatory, limitation of activity and/or home oxygen | 0 | 0 | 0
  Hospitalized Mild Disease, no oxygen therapy | 0 | 0 | 0
  Hospitalized Mild Disease, oxygen by mask or nasal prong | 34 | 40 | 74
  Hospitalized Severe Disease, humidified high-flow oxygen | 1 | 0 | 1
  Hospitalized Severe Disease, non-invasive ventilation | 0 | 0 | 0
  Hospitalized Severe Disease, intubation and mechanical ventilation | 0 | 0 | 0
  Hospitalized Severe Disease, ventilation + additional organ support-pressors, RRT, ECMO | 0 | 0 | 0
  Death | 0 | 0 | 0
NEWS2 [Median (Inter-Quartile Range); unit: units on a scale] — The National Early Warning Score 2 (NEWS2) has demonstrated an ability to discriminate patients at risk of poor outcomes. This score is based on 7 clinical parameters and ranges from 0 to 20. The NEWS2 is being used as an efficacy measure. Higher scores mean a worse outcome.
  units on a scale | 3 [3 to 5] | 4 [3 to 6] | 4 [3 to 6]
White Blood Cell (WBC) Count [Median (Inter-Quartile Range); unit: K cells/mcL] | 7.9 [5.6 to 10.8] | 6.8 [4.5 to 9.2] | 7.4 [5.1 to 10.4]
Neutrophil Count [Median (Inter-Quartile Range); unit: K cells/mcL] — Population: Lab test was not done for 2 participants in the Masked Saline Placebo group.
  K cells/mcL
    number analyzed (Participants) | 35 | 38 | 73
    (all) | 6.3 [3.8 to 8.8] | 5.7 [3.7 to 7.7] | 6 [3.7 to 8.4]
Total Lymphocyte Count [Median (Inter-Quartile Range); unit: K cells/mcL] — Population: Lab test was not done for 2 participants in the Masked Saline Placebo group.
  K cells/mcL
    number analyzed (Participants) | 35 | 38 | 73
    (all) | 0.9 [0.6 to 1.2] | 0.8 [0.6 to 1] | 0.9 [0.6 to 1.2]
Hemoglobin [Median (Inter-Quartile Range); unit: g/dL] | 13.5 [12.5 to 14.4] | 13.5 [11.4 to 14.1] | 13.5 [11.9 to 14.4]
Platelets [Median (Inter-Quartile Range); unit: K cells/mcL] | 246 [160 to 284] | 207 [137 to 294] | 229 [145 to 291]
Creatinine [Median (Inter-Quartile Range); unit: mg/dL] | 0.9 [0.78 to 1.2] | 1 [0.9 to 1.34] | 1 [0.83 to 1.23]
Glucose [Median (Inter-Quartile Range); unit: mg/dL] | 144 [120 to 206] | 160 [127 to 213] | 154 [124 to 206]
Alanine Transaminase (ALT/SGPT) [Median (Inter-Quartile Range); unit: U/L] — Population: Lab test was not done for 1 participant in the Convalescent Plasma group.
  U/L
    number analyzed (Participants) | 34 | 40 | 74
    (all) | 30 [21 to 52] | 31 [22 to 60] | 30 [21 to 59]
Aspartate Transaminase (AST/SGOT) [Median (Inter-Quartile Range); unit: U/L] — Population: Lab test was not done for 1 participant in the Convalescent Plasma group.
  U/L
    number analyzed (Participants) | 34 | 40 | 74
    (all) | 29 [24 to 47] | 35 [28 to 69] | 34 [25 to 49]
International Normalized Ratio (INR) [Median (Inter-Quartile Range); unit: unitless] — Population: Lab test was not done for 4 participants in the Convalescent Plasma group and 3 participants in the Masked Saline Placebo group.
  unitless
    number analyzed (Participants) | 31 | 37 | 68
    (all) | 1.11 [1.04 to 1.2] | 1.2 [1.1 to 1.3] | 1.15 [1.07 to 1.24]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Developing Acute Hypoxemic Respiratory Failure or All-cause Death
Description: Respiratory failure is defined as requiring mechanical ventilation, with or without endotracheal intubations, or extra-corporeal membrane oxygenation.
Time Frame: Day 1 through Day 28
Population: The primary outcome cannot be determined for 5 participants (4 in Convalescent Plasma, and 1 in Masked Saline Placebo) who terminated early from the study
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Masked Saline Placebo
Number analyzed (Participants) | 31 | 39
Participants | 3 | 4
Statistical Analysis 1: Comparison: Convalescent Plasma vs Masked Saline Placebo; Test type: Superiority; p = 1.00, Fisher Exact; Risk Difference (RD) = -0.01, 95% CI 2-sided [-0.15 to 0.14]

2. Secondary Outcome: Time (in Days) to Recovery
Description: Day of recovery is defined as the first day on which the subject satisfies one of the following three categories from the Modified World Health Organization (WHO) 8-point Ordinal Scale for Clinical Improvement : 1) Ambulatory, no limitation of activity; 2) Ambulatory, limitation of activity and/or home oxygen; 3) Hospitalized Mild Disease, no oxygen therapy.
Time Frame: Day 1 through Day 28
Population: All randomized participants are included in this analysis.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Convalescent Plasma | Masked Saline Placebo
Number analyzed (Participants) | 35 | 40
Days | 6 [4 to 9] | 6 [5 to 12.5]
Statistical Analysis 1: Comparison: Convalescent Plasma vs Masked Saline Placebo; Test type: Superiority; p = 0.749, Log Rank; Improvement Rate Ratio = 1.08, 95% CI 2-sided [0.65 to 1.78]

3. Secondary Outcome: Time (in Days) to Death or Respiratory Failure
Description: Defined as the first day on which the subject died from any cause or had respiratory failure. Respiratory failure is defined by requiring mechanical ventilation, with or without endotracheal intubations, or extra-corporeal membrane oxygenation.
Time Frame: Day 1 through Day 28
Population: All randomized participants are included in the analysis
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Convalescent Plasma | Masked Saline Placebo
Number analyzed (Participants) | 35 | 40
days | NA [NA to NA] — The median and inter-quartile range cannot be calculated because <25% of study participants experienced this event. | NA [NA to NA] — The median and inter-quartile range cannot be calculated because <25% of study participants experienced this event.
Statistical Analysis 1: Comparison: Convalescent Plasma vs Masked Saline Placebo; Test type: Superiority; p = 0.943, Log Rank; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.21 to 4.23]

4. Secondary Outcome: Proportion of Patients Who Died From Any Cause, Had Respiratory Failure, or Required Humidified Heated High-flow Nasal Cannula (HHHFNC) at >= 15 Lpm
Description: Defined as the proportion of subjects who died from any cause, had respiratory failure, or who required humidified heater high-flow cannula (HHHFNC) at >= 15 Lpm. Respiratory failure is defined by requiring mechanical ventilation, with or without endotracheal intubations, or extra-corporeal membrane oxygenation.
Time Frame: Day 1 through Day 28
Population: This secondary outcome cannot be determined for 5 participants (4 in Convalescent Plasma, and 1 in Masked Saline Placebo) who terminated early from the study
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Masked Saline Placebo
Number analyzed (Participants) | 31 | 39
Participants | 4 | 8
Statistical Analysis 1: Comparison: Convalescent Plasma vs Masked Saline Placebo; Test type: Superiority; p = 0.4014, Chi-squared; Risk Difference (RD) = -0.08, 95% CI 2-sided [-0.25 to 0.10]

5. Secondary Outcome: Time (in Days) to Death, Respiratory Failure, or HHHFNC at >= 15 Lpm
Description: Time to death or respiratory failure is defined as the first day on which the subject died from any cause, had respiratory failure (defined above), or who required HHHFNC at >= 15 Lpm.
Time Frame: Day 1 through Day 28
Population: All randomized participants were included in this analysis.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Convalescent Plasma | Masked Saline Placebo
Number analyzed (Participants) | 35 | 40
days | NA [NA to NA] — The median and inter-quartile range cannot be calculated because <25% of study participants experienced this event. | NA [NA to NA] — The median and inter-quartile range cannot be calculated because <25% of study participants experienced this event.
Statistical Analysis 1: Comparison: Convalescent Plasma vs Masked Saline Placebo; Test type: Superiority; p = 0.3762, Log Rank; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.18 to 1.96]

6. Secondary Outcome: Number of Participants With 28-day All-cause Mortality
Description: Death for Any Reason
Time Frame: Day 1 through Day 28
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Masked Saline Placebo
Number analyzed (Participants) | 31 | 39
Participants | 2 | 4
Statistical Analysis 1: Comparison: Convalescent Plasma vs Masked Saline Placebo; Test type: Superiority; p = 0.6867, Fisher Exact; Risk Difference (RD) = -0.04, 95% CI 2-sided [-0.17 to 0.09]

7. Secondary Outcome: Time to an Improvement of at Least One Category Using an Ordinal Scale
Description: Number of Days until the Modified WHO Clinical Status Improved by at Least One Category
  Modified WHO 8-point Ordinal Scale for Clinical Improvement. The scale is as follows: 0) No clinical or Virologic evidence of infection; 1) Ambulatory, no limitation of activity; 2) Ambulatory, limitation of activity and/or home oxygen; 3) Hospitalized Mild Disease, no oxygen therapy; 4) Hospitalized Mild Disease, oxygen by mask or nasal prong; 5a) Hospitalized Severe Disease, humidified high-flow oxygen; 5b) Hospitalized Severe Disease, non-invasive ventilation; 6) Hospitalized Severe Disease, intubation and mechanical ventilation; 7) Hospitalized Severe Disease, ventilation + additional organ support-pressors, renal replacement therapy (RRT), extracorporeal membrane oxygenation (ECMO); 8) Death. The higher the score, the worse the outcome.
Time Frame: Up through 28 days.
Population: All randomized participants were included in this analysis.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Convalescent Plasma | Masked Saline Placebo
Number analyzed (Participants) | 35 | 40
days | 6 [4 to 9] | 6 [5 to 12.5]
Statistical Analysis 1: Comparison: Convalescent Plasma vs Masked Saline Placebo; Test type: Superiority; p = 0.6494, Log Rank; Improvement Rate Ratio = 1.11, 95% CI 2-sided [0.68 to 1.83]

8. Secondary Outcome: Time to an Improvement of at Least Two Categories Using an Ordinal Scale
Description: Number of Days until the Modified WHO Clinical Status Improved by at Least Two Categories
  Modified WHO 8-point Ordinal Scale for Clinical Improvement. The scale is as follows: 0) No clinical or Virologic evidence of infection; 1) Ambulatory, no limitation of activity; 2) Ambulatory, limitation of activity and/or home oxygen; 3) Hospitalized Mild Disease, no oxygen therapy; 4) Hospitalized Mild Disease, oxygen by mask or nasal prong; 5a) Hospitalized Severe Disease, humidified high-flow oxygen; 5b) Hospitalized Severe Disease, non-invasive ventilation; 6) Hospitalized Severe Disease, intubation and mechanical ventilation; 7) Hospitalized Severe Disease, ventilation + additional organ support-pressors, RRT, ECMO; 8) Death. The higher the score, the worse the outcome.
Time Frame: Up through 28 days.
Population: All randomized participants were included in this analysis.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Convalescent Plasma | Masked Saline Placebo
Number analyzed (Participants) | 35 | 40
days | 7 [5 to 13] | 7 [5 to 16]
Statistical Analysis 1: Comparison: Convalescent Plasma vs Masked Saline Placebo; Test type: Superiority; p = 0.9338, Log Rank; Improvement Rate Ratio = 0.98, 95% CI 2-sided [0.59 to 1.63]

9. Secondary Outcome: Participant's Clinical Status by Ordinal Scale
Description: Modified WHO 8-point Ordinal Scale for Clinical Improvement. The scale is as follows: 0) No clinical or Virologic evidence of infection; 1) Ambulatory, no limitation of activity; 2) Ambulatory, limitation of activity and/or home oxygen; 3) Hospitalized Mild Disease, no oxygen therapy; 4) Hospitalized Mild Disease, oxygen by mask or nasal prong; 5a) Hospitalized Severe Disease, humidified high-flow oxygen; 5b) Hospitalized Severe Disease, non-invasive ventilation; 6) Hospitalized Severe Disease, intubation and mechanical ventilation; 7) Hospitalized Severe Disease, ventilation + additional organ support-pressors, RRT, ECMO; 8) Death. The higher the score, the worse the outcome.
Time Frame: Days 2, 4, 7, 11, 14, 21, and 28
Population: This secondary outcome cannot be determined for 3 participants (3 in Convalescent Plasma, and 0 in Masked Saline Placebo) who terminated on the day of randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Masked Saline Placebo
Number analyzed (Participants) | 32 | 40
Participants
  Day 2: Ambulatory, no limitation of activity | 0 | 0
  Day 2: Ambulatory, limitation of activity and/or home oxygen | 0 | 0
  Day 2: Hospitalized Mild Disease, no oxygen therapy | 1 | 1
  Day 2: Hospitalized Mild Disease, oxygen by mask or nasal prong | 28 | 35
  Day 2: Hospitalized Severe Disease, humidified high-flow oxygen | 1 | 3
  Day 2: Hospitalized Severe Disease, non-invasive ventilation | 2 | 0
  Day 2: Hospitalized Severe Disease, intubation and mechanical ventilation | 0 | 0
  Day 2: Hospitalized Severe Disease, ventilation + additional organ support-pressors, RRT, ECMO | 0 | 1
  Day 2: Death | 0 | 0
  Day 4: Ambulatory, no limitation of activity | 2 | 2
  Day 4: Ambulatory, limitation of activity and/or home oxygen | 2 | 6
  Day 4: Hospitalized Mild Disease, no oxygen therapy | 6 | 1
  Day 4: Hospitalized Mild Disease, oxygen by mask or nasal prong | 19 | 23
  Day 4: Hospitalized Severe Disease, humidified high-flow oxygen | 1 | 6
  Day 4: Hospitalized Severe Disease, non-invasive ventilation | 0 | 0
  Day 4: Hospitalized Severe Disease, intubation and mechanical ventilation | 1 | 1
  Day 4: Hospitalized Severe Disease, ventilation + additional organ support-pressors, RRT, ECMO | 1 | 1
  Day 4: Death | 0 | 0
  Day 7: number analyzed (Participants) | 30 | 39
  Day 7: Ambulatory, no limitation of activity | 6 | 4
  Day 7: Ambulatory, limitation of activity and/or home oxygen | 11 | 17
  Day 7: Hospitalized Mild Disease, no oxygen therapy | 2 | 3
  Day 7: Hospitalized Mild Disease, oxygen by mask or nasal prong | 8 | 10
  Day 7: Hospitalized Severe Disease, humidified high-flow oxygen | 2 | 3
  Day 7: Hospitalized Severe Disease, non-invasive ventilation | 0 | 0
  Day 7: Hospitalized Severe Disease, intubation and mechanical ventilation | 1 | 1
  Day 7: Hospitalized Severe Disease, ventilation + additional organ support-pressors, RRT, ECMO | 0 | 1
  Day 7: Death | 0 | 0
  Day 11: number analyzed (Participants) | 30 | 38
  Day 11: Ambulatory, no limitation of activity | 5 | 5
  Day 11: Ambulatory, limitation of activity and/or home oxygen | 17 | 23
  Day 11: Hospitalized Mild Disease, no oxygen therapy | 3 | 1
  Day 11: Hospitalized Mild Disease, oxygen by mask or nasal prong | 2 | 6
  Day 11: Hospitalized Severe Disease, humidified high-flow oxygen | 2 | 1
  Day 11: Hospitalized Severe Disease, non-invasive ventilation | 0 | 0
  Day 11: Hospitalized Severe Disease, intubation and mechanical ventilation | 1 | 0
  Day 11: Hospitalized Severe Disease, ventilation + additional organ support-pressors, RRT, ECMO | 0 | 1
  Day 11: Death | 0 | 1
  Day 14: number analyzed (Participants) | 29 | 36
  Day 14: Ambulatory, no limitation of activity | 6 | 5
  Day 14: Ambulatory, limitation of activity and/or home oxygen | 18 | 23
  Day 14: Hospitalized Mild Disease, no oxygen therapy | 2 | 2
  Day 14: Hospitalized Mild Disease, oxygen by mask or nasal prong | 2 | 5
  Day 14: Hospitalized Severe Disease, humidified high-flow oxygen | 0 | 1
  Day 14: Hospitalized Severe Disease, non-invasive ventilation | 0 | 0
  Day 14: Hospitalized Severe Disease, intubation and mechanical ventilation | 1 | 0
  Day 14: Hospitalized Severe Disease, ventilation + additional organ support-pressors, RRT, ECMO | 0 | 0
  Day 14: Death | 0 | 0
  Day 21: number analyzed (Participants) | 29 | 36
  Day 21: Ambulatory, no limitation of activity | 7 | 9
  Day 21: Ambulatory, limitation of activity and/or home oxygen | 16 | 24
  Day 21: Hospitalized Mild Disease, no oxygen therapy | 3 | 1
  Day 21: Hospitalized Mild Disease, oxygen by mask or nasal prong | 2 | 2
  Day 21: Hospitalized Severe Disease, humidified high-flow oxygen | 0 | 0
  Day 21: Hospitalized Severe Disease, non-invasive ventilation | 0 | 0
  Day 21: Hospitalized Severe Disease, intubation and mechanical ventilation | 1 | 0
  Day 21: Hospitalized Severe Disease, ventilation + additional organ support-pressors, RRT, ECMO | 0 | 0
  Day 21: Death | 0 | 0
  Day 28: number analyzed (Participants) | 29 | 35
  Day 28: Ambulatory, no limitation of activity | 6 | 11
  Day 28: Ambulatory, limitation of activity and/or home oxygen | 20 | 23
  Day 28: Hospitalized Mild Disease, no oxygen therapy | 0 | 0
  Day 28: Hospitalized Mild Disease, oxygen by mask or nasal prong | 3 | 1
  Day 28: Hospitalized Severe Disease, humidified high-flow oxygen | 0 | 0
  Day 28: Hospitalized Severe Disease, non-invasive ventilation | 0 | 0
  Day 28: Hospitalized Severe Disease, intubation and mechanical ventilation | 0 | 0
  Day 28: Hospitalized Severe Disease, ventilation + additional organ support-pressors, RRT, ECMO | 0 | 0
  Day 28: Death | 0 | 0

10. Secondary Outcome: Change in the Ordinal Scale From Baseline to Days 2, 4, 7, 11, 14, 21, and 28
Description: Change in the Modified WHO Clinical Status
  Modified WHO 8-point Ordinal Scale for Clinical Improvement. The scale is as follows: 0) No clinical or Virologic evidence of infection; 1) Ambulatory, no limitation of activity; 2) Ambulatory, limitation of activity and/or home oxygen; 3) Hospitalized Mild Disease, no oxygen therapy; 4) Hospitalized Mild Disease, oxygen by mask or nasal prong; 5a) Hospitalized Severe Disease, humidified high-flow oxygen; 5b) Hospitalized Severe Disease, non-invasive ventilation; 6) Hospitalized Severe Disease, intubation and mechanical ventilation; 7) Hospitalized Severe Disease, ventilation + additional organ support-pressors, RRT, ECMO; 8) Death. The higher the score, the worse the outcome.
Time Frame: From Baseline to Days 2, 4, 7, 11, 14, 21, and 28.
Population: as for outcome 9
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Convalescent Plasma | Masked Saline Placebo
Number analyzed (Participants) | 32 | 40
units on a scale
  Baseline to Day 2 | 0 [-1 to 1] | 0 [-1 to 3]
  Baseline to Day 4 | 0 [-3 to 3] | 0 [-3 to 3]
  Baseline to Day 7: number analyzed (Participants) | 30 | 39
  Baseline to Day 7 | -2 [-3 to 1] | -2 [-3 to 3]
  Baseline to Day 11: number analyzed (Participants) | 30 | 38
  Baseline to Day 11 | -2 [-3 to 1] | -2 [-3 to 4]
  Baseline to Day 14: number analyzed (Participants) | 29 | 36
  Baseline to Day 14 | -2 [-3 to 1] | -2 [-3 to 1]
  Baseline to Day 21: number analyzed (Participants) | 29 | 36
  Baseline to Day 21 | -2 [-3 to 1] | -2 [-3 to 0]
  Baseline to Day 28: number analyzed (Participants) | 29 | 35
  Baseline to Day 28 | -2 [-3 to 0] | -2 [-3 to 0]

11. Secondary Outcome: Categorical Change in the Ordinal Scale From Baseline to Days 2, 4, 7, 11, 14, 21, and 28
Description: Categorical Change in the Modified WHO 8-point Ordinal Scale for Clinical Improvement
  Modified WHO 8-point Ordinal Scale for Clinical Improvement. The scale is as follows: 0) No clinical or Virologic evidence of infection; 1) Ambulatory, no limitation of activity; 2) Ambulatory, limitation of activity and/or home oxygen; 3) Hospitalized Mild Disease, no oxygen therapy; 4) Hospitalized Mild Disease, oxygen by mask or nasal prong; 5a) Hospitalized Severe Disease, humidified high-flow oxygen; 5b) Hospitalized Severe Disease, non-invasive ventilation; 6) Hospitalized Severe Disease, intubation and mechanical ventilation; 7) Hospitalized Severe Disease, ventilation + additional organ support-pressors, RRT, ECMO; 8) Death. The higher the score, the worse the outcome.
Time Frame: From Baseline to Days 2, 4, 7, 11, 14, 21, and 28.
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Masked Saline Placebo
Number analyzed (Participants) | 32 | 40
Participants
  Baseline to Day 2: 4 Point Improvement | 0 | 0
  Baseline to Day 2: 3 Point Improvement | 0 | 0
  Baseline to Day 2: 2 Point Improvement | 0 | 0
  Baseline to Day 2: 1 Point Improvement | 1 | 1
  Baseline to Day 2: No Change | 29 | 35
  Baseline to Day 2: 1 Point Worsening | 2 | 3
  Baseline to Day 2: 2 Point Worsening | 0 | 0
  Baseline to Day 2: 3 Point Worsening | 0 | 1
  Baseline to Day 2: 4 Point Worsening | 0 | 0
  Baseline to Day 4: 4 Point Improvement | 0 | 0
  Baseline to Day 4: 3 Point Improvement | 2 | 2
  Baseline to Day 4: 2 Point Improvement | 2 | 6
  Baseline to Day 4: 1 Point Improvement | 6 | 1
  Baseline to Day 4: No Change | 19 | 23
  Baseline to Day 4: 1 Point Worsening | 2 | 6
  Baseline to Day 4: 2 Point Worsening | 0 | 1
  Baseline to Day 4: 3 Point Worsening | 1 | 1
  Baseline to Day 4: 4 Point Worsening | 0 | 0
  Baseline to Day 7: number analyzed (Participants) | 30 | 39
  Baseline to Day 7: 4 Point Improvement | 0 | 0
  Baseline to Day 7: 3 Point Improvement | 6 | 4
  Baseline to Day 7: 2 Point Improvement | 11 | 17
  Baseline to Day 7: 1 Point Improvement | 2 | 3
  Baseline to Day 7: No Change | 8 | 10
  Baseline to Day 7: 1 Point Worsening | 3 | 3
  Baseline to Day 7: 2 Point Worsening | 0 | 1
  Baseline to Day 7: 3 Point Worsening | 0 | 1
  Baseline to Day 7: 4 Point Worsening | 0 | 0
  Baseline to Day 11: number analyzed (Participants) | 30 | 38
  Baseline to Day 11: 4 Point Improvement | 0 | 0
  Baseline to Day 11: 3 Point Improvement | 5 | 5
  Baseline to Day 11: 2 Point Improvement | 17 | 23
  Baseline to Day 11: 1 Point Improvement | 3 | 1
  Baseline to Day 11: No Change | 2 | 6
  Baseline to Day 11: 1 Point Worsening | 3 | 1
  Baseline to Day 11: 2 Point Worsening | 0 | 0
  Baseline to Day 11: 3 Point Worsening | 0 | 1
  Baseline to Day 11: 4 Point Worsening | 0 | 1
  Baseline to Day 14: number analyzed (Participants) | 29 | 36
  Baseline to Day 14: 4 Point Improvement | 0 | 0
  Baseline to Day 14: 3 Point Improvement | 6 | 5
  Baseline to Day 14: 2 Point Improvement | 18 | 23
  Baseline to Day 14: 1 Point Improvement | 2 | 2
  Baseline to Day 14: No Change | 2 | 5
  Baseline to Day 14: 1 Point Worsening | 1 | 1
  Baseline to Day 14: 2 Point Worsening | 0 | 0
  Baseline to Day 14: 3 Point Worsening | 0 | 0
  Baseline to Day 14: 4 Point Worsening | 0 | 0
  Baseline to Day 21: number analyzed (Participants) | 29 | 36
  Baseline to Day 21: 4 Point Improvement | 0 | 0
  Baseline to Day 21: 3 Point Improvement | 7 | 9
  Baseline to Day 21: 2 Point Improvement | 16 | 24
  Baseline to Day 21: 1 Point Improvement | 3 | 1
  Baseline to Day 21: No Change | 2 | 2
  Baseline to Day 21: 1 Point Worsening | 1 | 0
  Baseline to Day 21: 2 Point Worsening | 0 | 0
  Baseline to Day 21: 3 Point Worsening | 0 | 0
  Baseline to Day 21: 4 Point Worsening | 0 | 0
  Baseline to Day 28: number analyzed (Participants) | 29 | 35
  Baseline to Day 28: 4 Point Improvement | 0 | 0
  Baseline to Day 28: 3 Point Improvement | 6 | 11
  Baseline to Day 28: 2 Point Improvement | 20 | 23
  Baseline to Day 28: 1 Point Improvement | 1 | 0
  Baseline to Day 28: No Change | 2 | 1
  Baseline to Day 28: 1 Point Worsening | 0 | 0
  Baseline to Day 28: 2 Point Worsening | 0 | 0
  Baseline to Day 28: 3 Point Worsening | 0 | 0
  Baseline to Day 28: 4 Point Worsening | 0 | 0

12. Secondary Outcome: Time to Discharge or to a National Early Warning Score 2 (NEWS2) of <= 2 Maintained for at Least 22 Hours, Whichever Occurs First
Description: Number of Days until Initial Hospitalization Discharge or (NEWS2 <= 2 Maintained for at Least 22 Hours)
  The National Early Warning Score 2 (NEWS2) score has demonstrated an ability to discriminate patients at risk of poor outcomes. This score is based on 7 clinical parameters and ranges from 0 to 20. The NEWS2 is being used as an efficacy measure. Higher scores mean a worse outcome.
Time Frame: Up through 28 days.
Population: All randomized participants were included in this analysis.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Convalescent Plasma | Masked Saline Placebo
Number analyzed (Participants) | 35 | 40
days | 4 [3 to 7] | 4.5 [3 to 10.5]
Statistical Analysis 1: Comparison: Convalescent Plasma vs Masked Saline Placebo; Test type: Superiority; p = 0.5682, Log Rank; Improvement Rate Ratio = 1.14, 95% CI 2-sided [0.70 to 1.86]

13. Secondary Outcome: Change in National Early Warning Score 2 (NEWS2) From Day 1 (Baseline) to Days 2, 4, 7, 11, 15, and 29
Description: Change in NEWS2
  The National Early Warning Score 2 (NEWS2) has demonstrated an ability to discriminate patients at risk of poor outcomes. This score is based on 7 clinical parameters and ranges from 0 to 20. The NEWS2 is being used as an efficacy measure. Higher scores mean a worse outcome.
Time Frame: From Day 1 (baseline) to Days 2, 4, 7, 11, 15, and 29
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Convalescent Plasma | Masked Saline Placebo
Number analyzed (Participants) | 32 | 40
score on a scale
  Day 1 to Day 2 | 0 [-0.5 to 1] | 0 [-1 to 1]
  Day 1 to Day 4: number analyzed (Participants) | 28 | 32
  Day 1 to Day 4 | -0.5 [-2 to 1] | -1 [-2 to 1]
  Day 1 to Day 7: number analyzed (Participants) | 13 | 17
  Day 1 to Day 7 | -1 [-2 to 0] | 0 [-3 to 2]
  Day 1 to Day 11: number analyzed (Participants) | 8 | 10
  Day 1 to Day 11 | -2 [-3 to -0.5] | -1 [-1 to 0]
  Day 1 to Day 15: number analyzed (Participants) | 11 | 20
  Day 1 to Day 15 | -2 [-3 to -1] | -1.5 [-3 to -1]
  Day 1 to Day 29: number analyzed (Participants) | 18 | 19
  Day 1 to Day 29 | -2 [-3 to -2] | -2 [-5 to -1]

14. Secondary Outcome: Duration of Hospitalization
Description: Number of Days Hospitalized During Initial Hospitalization
Time Frame: Day 1 through Day 28
Population: This secondary outcome cannot be determined for 3 participants (3 in Convalescent Plasma, and 0 in Masked Saline Placebo) who terminated early on the day of randomization.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Convalescent Plasma | Masked Saline Placebo
Number analyzed (Participants) | 32 | 40
days | 5.5 [4 to 8.5] | 6 [4 to 10.5]
Statistical Analysis 1: Comparison: Convalescent Plasma vs Masked Saline Placebo; Test type: Superiority; p = 0.8642, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-2.3 to 2.3]

15. Secondary Outcome: Incidence of Discontinuation or Temporary Suspension of Study Product Administrations (for Any Reason)
Description: Number of participants for whom study product administration was discontinued or temporarily suspended for any reason
Time Frame: Day 1 through Day 3
Population: 3 participants in the Convalescent Plasma group withdrew from the study prior to study product administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Masked Saline Placebo
Number analyzed (Participants) | 32 | 40
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 days
Description: The study requires reporting of the following types of events :
  1. All serious adverse events,
  2. Treatment-related adverse events at any severity, and
  3. All grade 3 adverse events regardless of relatedness to study product.
Arm/Group | Convalescent Plasma | Masked Saline Placebo
All-Cause Mortality (participants affected / at risk) | 3/35 | 4/40
Serious Adverse Events (participants affected / at risk) | 8/35 | 5/40
Other Adverse Events (participants affected / at risk) | 5/35 | 9/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Convalescent Plasma (N=35) | Masked Saline Placebo (N=40)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
COVID-19 Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Diabetic Foot Infection (Infections and infestations) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Electrocardiogram ST Segment Elevation (Investigations) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Convalescent Plasma (N=35) | Masked Saline Placebo (N=40)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Oxygen Consumption Increased (Investigations) | 1 (1) | 4 (4)
Fluid Overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Intensive Care (Surgical and medical procedures) | 1 (1) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive Urgency (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT04539275/Prot_SAP_001.pdf
  • Informed Consent Form (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT04539275/ICF_000.pdf